CLINICAL TRIAL: NCT03906201
Title: Effect of Phytoecdysterone Administration on Cytotoxicity, Genotoxicity and Metabolic Control in Subjects With Prediabetes
Brief Title: Effect of Phytoecdysterone Administration in Subjects With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Ana Lilia Fletes Rayas, Reseach Professor Associated, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 125/18
Record Dates: First submitted 2018-09-11; First posted 2019-04-08 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: PreDiabetes
Keywords: PreDiabetes; Ecdysterone; Genotoxicity; Citotoxicity; Micronuclei; Glycemic Control
MeSH Terms: conditions — Prediabetic State | interventions — Ecdysterone

STUDY DESIGN:
Intervention Model Description: cohort populations with diagnostic metabolic syndrome treatment base with ecdysterone for 90 days
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Randomized double-blind clinical trial plus control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Subjects diagnosed with prediabetes according to the criteria of the American Diabetes Association, version 2019 with placebo treatment
  Interventions: Other: Placebo
- Ecdysterone Group (Experimental): Subjects diagnosed with prediabetes according to the criteria of the American Diabetes Association, version 2019 whit ecdysterone treatment
  Interventions: Dietary Supplement: Ecdysterone

INTERVENTIONS:
Dietary Supplement: Ecdysterone — Food supplement of plant origin with pronounced biological activity and potentially hypoglycaemic
  Arms: Ecdysterone Group
Other: Placebo — no pharmacologic effect
  Other Names: magnesia stearate
  Arms: Control Group

SUMMARY:
Prediabetes is the term used for people whose glucose levels do not meet the criteria for diabetes but are too high to be considered normal. This is defined by the presence of blood glucose between 100-125 mg / dL, values per glucose tolerance curve of 140-199mg / dL and/or HbA1c 5.7-6.4%. Prediabetes should not be considered as a clinical entity in itself, but as a risk factor for diabetes and cardiovascular disease (CVD). Prediabetes is associated with obesity (especially abdominal or visceral obesity), dyslipidemia with elevated triglycerides and/or low HDL cholesterol, and hypertension.

DETAILED DESCRIPTION:
Subjects with a diagnosis of prediabetes are included according to the criteria of the American Diabetes Association in its version 2019, between 30 and 60 years old residents of the city of Guadalajara, Jalisco, Mexico who come to clinical nutrition consultation in the University Hospital Fray Antonio Alcalde from the city of Guadalajara, Jalisco, Mexico.

The study design is a randomized, randomized clinical trial with a control group in two groups: an intervention group with ecdysterone 300mg every 24 hours for 12 weeks (approximately 90 days) and an approved placebo control group (magnesia stearate) ) at 300mg every 24 hours for 12 weeks (approximately 90 days).

ELIGIBILITY:
Inclusion Criteria:

1. - Fasting Plasma Glucose between 100 mg/dL (5.6 mmol/L) to 125 mg/dL (6.9 mmol/L)
2. - Oral Glucose Tolerance Test 140 mg/dL (7.8 mmol/L) to 199 mg/dL (11.0 mmol/L)
3. - A1C 5.7-6.4% (39-47 mmol/mol).
4. - Body Mass Index >25 kg/m2 or >23 kg/m2
5. - Adults who have one or more of the following risk factors:

   * First-degree relative with diabetes
   * High-risk race/ethnicity
   * History of CVD
6. - Blood Pressure <140/90 mmHg without therapy for hypertension
7. - HDL cholesterol level <0.35 mg/dL (0.90 mmol/L) and/or a triglyceride level >0.250 mg/dL (2.82 mmol/L)

Exclusion Criteria:

1.- Pregnant women or lactic period 2- Patients with some other chronic degenerative disease like diabetes mellitus 2 with pharmacologic treatment.

3.- Hypertension 4.- Cancer, 5.- Hyperthyroidism 6.- Hypothyroidism 7.- Immunologic disease 8.- Kidney disease 9.- Hepatic disease 10.- Cardiovascular disease 11- Abaqus activity 12.-Alcoholic activity.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the number of micronuclei after 90 days | 90 days
  The number of micronuclei will be evaluated at baseline and day 90 with Schmidt technique by giemsa/wright and the entered values reflect the number of micronuceli at day 90
Changes in fasting glucose levels after 90 days of intervention with betaecdysterone and placebo | 90 days
  The fasting glucose levels will be evaluated at baseline and day 90 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at day 90
Changes in glycosylated hemoglobin (A1C) after 90 days of intervention with betaecdysterone and placebo | 90 days
  Glycosylated hemoglobin will be evaluated at baseline and day 90 by high pressure liquid chromatography (HPLC) and the entered values reflect the glycosylated hemoglobin at day 90

SECONDARY OUTCOMES:
Body Weight | 90 days
  The body weight will be measured at baseline, day 30, day 60 and day 90 with a bioimpedance balance and the entered values reflect the body weight at 90 days
Body Mass Index | 90 days
  Body Mass Index will be calculated at baseline, day 30, day 60 and day 90 with the Quetelet index formula and the entered values reflect the body mass index at day 90
Waist Circumference | 90 days
  Waist circumference will be evaluated at baseline and at day 90 with a flexible tape
Total Cholesterol | 90 days
  Total cholesterol levels will be evaluated at baseline and day 90 by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at day 90
Triglycerides levels | 90 days
  Triglycerides levels will be evaluated at baseline and day 90 with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at day 90
High Density Lipoprotein (c-HDL) levels | 90 days
  c-HDL levels will be evaluated at baseline and day 90 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at day 90
Low Density Lipoproteins (c-LDL) levels | 90 days
  c-LDL levels will be evaluated at baseline and day 90 with enzymatic/colorimetric techniques and the entered values reflect the c-LDL level at day 90
Creatinine levels | 90 days
  Creatinine levels will be evaluated at baseline and day 90 with enzymatic/colorimetric techniques
Alanine aminotransferase (ALT) levels | 90 days
  ALT levels will be evaluated at baseline and day 90 with enzymatic/colorimetric techniques
Aspartate aminotransferase (AST) levels | 90 days
  AST levels will be evaluated at baseline and day 90 enzymatic/colorimetric techniques
Blood pressure | 90 days
  Blood pressure will be measured at baseline and day 90 with a digital sphygmomanometer and the entered values reflect the blood pressure at day 90

CONTACTS AND LOCATIONS:
Overall Officials: ANA FLETES, Principal Investigator — University of Guadalajara
Locations (1):
- Ana Fletes, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
THE RESULTS GENERATED AND THE PERSONAL DATA OF THE PARTICIPANTS ARE ON THE CONSENT OF THE SUBJECT OF STUDY AND OF THE PRINCIPAL INVESTIGATOR. THEY ARE EXTRICTLY CONFIDENTIAL AND WILL ONLY BE USED BY HOSPITAL DOCTORS

REFERENCES:
- [Background] Álvarez-Gasca Ma, Hernández-Pozo MR, Jiménez-Martínez M, Durán-Díaz A. Estilo de vida y presencia de síndrome metabólico en estudiantes universitarios. Diferencias por sexo. Rev de psicología. 2014; 32(1):121-138
- [Background] Andreassi MG, Barale R, Iozzo P, Picano E. The association of micronucleus frequency with obesity, diabetes and cardiovascular disease. Mutagenesis. 2011 Jan;26(1):77-83. doi: 10.1093/mutage/geq077. PMID 21164186
- [Background] •Aparicio MR, Estrada LA, Fernández C, Hernández RM, Ruiz M, Ramos D, et al. Manual de antropometría. Instituto nacional de ciencias médicas y nutrición salvador zubirán: 2014 citar en:http://www.facmed.unam.mx/deptos/salud/censenanza/spi/unidad2/antropometria_manualinnsz.pdf
- [Background] Berti C, Riso P, Monti LD, Porrini M. In vitro starch digestibility and in vivo glucose response of gluten-free foods and their gluten counterparts. Eur J Nutr. 2004 Aug;43(4):198-204. doi: 10.1007/s00394-004-0459-1. Epub 2004 Jan 6. PMID 15309439
- [Background] Graf BL, Poulev A, Kuhn P, Grace MH, Lila MA, Raskin I. Quinoa seeds leach phytoecdysteroids and other compounds with anti-diabetic properties. Food Chem. 2014 Nov 15;163:178-85. doi: 10.1016/j.foodchem.2014.04.088. Epub 2014 May 4. PMID 24912714
- [Background] FAO, 2013. Food and agriculture organization of the united nations rome. Http://www.fao.org/docrep/018/i3300e/i3300e00.pdf
- [Background] FAO. Food and agriculture organization of the united nations 2011. La quinua: cultivo milenario para contribuir a la seguridad alimentaria mundial. Http://www.fao.org/docrep/017/aq287s/aq287s.pdf
- [Background] Figuerola F, Muñoz O, Estévez AM. La linaza como fuente de compuestos bioactivos para la elaboración de alimentos. Agro sur. 2008; 36(2): 49-58. Doi:10.4206/agrosur.2008.v36n2-01
- [Background] Gutiérrez JP, Rivera-Dommarco J, Shamah-Levy T, Villalpando-Hernández S, Franco A, Cuevas-Nasu l, et al. Encuesta nacional de salud y nutrición 2012. Resultados nacionales. Cuernavaca, méxico: instituto nacional de salud pública (mx), 2012
- [Background] Harishankar MK, Logeshwaran S, Sujeevan S, Aruljothi KN, Dannie MA, Devi A. Genotoxicity evaluation of metformin and glimepiride by micronucleus assay in exfoliated urothelial cells of type 2 diabetes mellitus patients. Food Chem Toxicol. 2015 Sep;83:146-50. doi: 10.1016/j.fct.2015.06.013. Epub 2015 Jun 24. PMID 26115598
- [Background] Karaman A, Aydin H, Geckinli B, Cetinkaya A, Karaman S. DNA damage is increased in lymphocytes of patients with metabolic syndrome. Mutat Res Genet Toxicol Environ Mutagen. 2015 Apr;782:30-5. doi: 10.1016/j.mrgentox.2015.03.009. Epub 2015 Mar 13. PMID 25868129
- [Background] Leon-Munoz LM, Guallar-Castillon P, Lopez Garcia E, Banegas JR, Gutierrez-Fisac JL, Rodriguez-Artalejo F. Relationship of BMI, waist circumference, and weight change with use of health services by older adults. Obes Res. 2005 Aug;13(8):1398-404. doi: 10.1038/oby.2005.169. PMID 16129722
- [Background] Lizarzaburu-Robles JC. Síndrome metabólico: metabolicsyndrome: concept and practical application. An facmed. 2013;74(4):315-320.
- [Background] Kaufer-Horwitz M, Toussaint G. Indicadores antropométricos para evaluar sobrepeso y obesidad en pediatría. Bol. Med. Hosp. Infant. Mex; 2008;65(6): 502-518.
- [Background] Moreno-Altamirano l, García-García JJ, Soto-Estrada G, Capraro S, Limón-Cruz D. Epidemiología y determinantes sociales asociados a la obesidad y la diabetes tipo 2 en méxico. Revmedhosp gen méx. 2014; 77(3):86-95.
- [Background] Morris D, Vaisey-Genserb. Availability and labeling of flaxseedfood, products and supplements. In: thompson, l. U.; cunnane s. C. Flaxseed in human nutrition. 2003. 2nd edn., champaign, illinois. Aocs press. Pp. 404-422.
- [Background] Murakami A, Ashida H, Terao J. Multitargeted cancer prevention by quercetin. Cancer Lett. 2008 Oct 8;269(2):315-25. doi: 10.1016/j.canlet.2008.03.046. Epub 2008 May 7. PMID 18467024
- [Background] Ojeda-Lavin A. Proyecciones de la población 2010-2050. Consejo nacional de población méxico. 2014.http://www.conapo.gob.mx/es/conapo/proyecciones.
- [Background] Omsa. Datos y cifras. 10 datos sobre la obesidad. 2015. Disponible en: http://www.who.int/features/factfiles/obesity/facts/es/index1.html
- [Background] Cuevas ZO, Sangronis E. [Characterization of flaxseed (Linum usitatissimum L.) grown in Venezuela]. Arch Latinoam Nutr. 2012 Jun;62(2):192-200. Spanish. PMID 23610908
- [Background] Penarrieta JM, Alvarado JA, Akesson B, Bergenstahl B. Total antioxidant capacity and content of flavonoids and other phenolic compounds in canihua (Chenopodium pallidicaule): an Andean pseudocereal. Mol Nutr Food Res. 2008 Jun;52(6):708-17. doi: 10.1002/mnfr.200700189. PMID 18537130
- [Background] Rajesha J, Murthy KN, Kumar MK, Madhusudhan B, Ravishankar GA. Antioxidant potentials of flaxseed by in vivo model. J Agric Food Chem. 2006 May 31;54(11):3794-9. doi: 10.1021/jf053048a. PMID 16719498
- [Background] Ramcharitar A, Badrie N, Mattfeldtbeman M, Matsuo H, Ridley C. Consumeracceptability of muffinswithflaxseed (linumusitatissimum). J. Foodsci 2005;70: 504-507.
- [Background] Ranilla LG, Apostolidis E, Genovese MI, Lajolo FM, Shetty K. Evaluation of indigenous grains from the Peruvian Andean region for antidiabetes and antihypertension potential using in vitro methods. J Med Food. 2009 Aug;12(4):704-13. doi: 10.1089/jmf.2008.0122. PMID 19735168
- [Background] Repo-Carrasco-Valencia R, Hellströmb JK, Juha-Matti P, Mattila PH. Flavonoids and other phenolic compounds in andean indigenous grains: quinoa (chenopodium quinoa), kañiwa (chenopodium pallidicaule) and kiwicha (amaranthus caudatus). Food chemistry. 2010; 120(1):128-133.
- [Background] Shahidi F, Kim SK. Quality management of marine nutraceuticals. In: ho c-t, zheng qy, editors. Quality management of nutraceuticals. Acs symposium series 803. Washington, d.c.: american chemical society. 2002.p. 76-87.
- [Background] Spedding G, Ratty A, Middleton E Jr. Inhibition of reverse transcriptases by flavonoids. Antiviral Res. 1989 Sep;12(2):99-110. doi: 10.1016/0166-3542(89)90073-9. PMID 2480745
- [Background] Stewart LK, Soileau JL, Ribnicky D, Wang ZQ, Raskin I, Poulev A, Majewski M, Cefalu WT, Gettys TW. Quercetin transiently increases energy expenditure but persistently decreases circulating markers of inflammation in C57BL/6J mice fed a high-fat diet. Metabolism. 2008 Jul;57(7 Suppl 1):S39-46. doi: 10.1016/j.metabol.2008.03.003. PMID 18555853
- [Background] Torres-Bugarín O, Ramos-Ibarra ML. Utilidad de la prueba de micronúcleos y anormalidades nucleares en células exfoliadas de mucosa oral en la evaluación de daño genotóxico y citotóxico. Int. J. Morphol. 2013. 31(2):650-657.
- [Background] Torres-Bugarín O, Zavala-cerna MG, Macriz-Romero N, Flores-García A, Ramos-Ibarra ML. Procedimientos básicos de la prueba de micronúcleos y anormalidades nucleares en células exfoliadas de mucosa oral. El residente. 2013; (8):4-11.
- [Background] Voss S, Hesse A, Zimmermann DJ, Sauerbruch T, von Unruh GE. Intestinal oxalate absorption is higher in idiopathic calcium oxalate stone formers than in healthy controls: measurements with the [(13)C2]oxalate absorption test. J Urol. 2006 May;175(5):1711-5. doi: 10.1016/S0022-5347(05)01001-3. PMID 16600737
- [Background] Hou Y, Aboukhatwa MA, Lei DL, Manaye K, Khan I, Luo Y. Anti-depressant natural flavonols modulate BDNF and beta amyloid in neurons and hippocampus of double TgAD mice. Neuropharmacology. 2010 May;58(6):911-20. doi: 10.1016/j.neuropharm.2009.11.002. Epub 2009 Nov 14. PMID 19917299
- [Background] Zimmet P, M M Alberti KG, Serrano Rios M. [A new international diabetes federation worldwide definition of the metabolic syndrome: the rationale and the results]. Rev Esp Cardiol. 2005 Dec;58(12):1371-6. No abstract available. Spanish. PMID 16371194
- [Background] Zong G, Demark-Wahnefried W, Wu H, Lin X. Effects of flaxseed supplementation on erythrocyte fatty acids and multiple cardiometabolic biomarkers among Chinese with risk factors of metabolic syndrome. Eur J Nutr. 2013 Aug;52(5):1547-51. doi: 10.1007/s00394-012-0461-y. Epub 2012 Nov 23. PMID 23179200
- See also: The journal of clinical and applied research and education. Diabetes Care. American Diabetes Association. Standards of Medical Care in Diabetes-2019. — http://fmdiabetes.org/wp-content/uploads/2019/01/ada-2019.pdf